CLINICAL TRIAL: NCT06531226
Title: Personality Traits and Colonoscopy Insertion Time: Applying Machine Learning to Predict the Colonoscopy Time and Difficult Colonoscopy
Brief Title: Difficult Colonoscopy and Personality Traits
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202406-030
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Disorders
Keywords: machine learning; difficult colonoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High neuroticism score group: The neuroticism score was higher than the average score identified by the norm
  Interventions: Other: Fill in personality questionnaires
- Low neuroticism score group: The neuroticism score was lower than the average score identified by the norm
  Interventions: Other: Fill in personality questionnaires

INTERVENTIONS:
Other: Fill in personality questionnaires — For patients who need to undergo colonoscopy, we invite them to fill out a personality survey questionnaire after obtaining their informed consent. The questionnaire contains 60 survey questions, which cover the five dimensions of the Big Five personality traits. Each question has five options, corresponding to the five states of very disagree to very agree. The questionnaire was developed based on the Chinese population and has four norms applicable to different age groups to ensure the reliability of the questionnaire.

SUMMARY:
The cecal intubation time (CIT) refers to the time required for the tip of the colonoscope to reach the cecum from passing through the anus. A prolonged CIT is considered a marker of difficulty in colonoscopy. CIT greater than 10 minutes is considered a difficult colonoscopy. Studies have identified factors that influence CIT, including age, gender, body mass index (BMI), waist circumference, bowel preparation, prior abdominal surgery, etc. Personality traits have been found to be associated with the onset of many diseases, such as hypertension and A-type personality, depression and neurotic personality. According to the Big Five personality theory, personality can be decomposed into five dimensions: openness (O), conscientiousness (C), extraversion (E), agreeableness (A), and neuroticism (N). There is a lack of research on the association between personality traits and colonoscopy insertion time, and the purpose of this study is to investigate whether personality, BMI, age, gender, anxiety and depression index, metabolic diseases, and abdominal pelvic surgery history lead to prolonged colonoscopy insertion time and difficult colonoscopy, and to identify significant variables as predictors by using machine learning methods to build a clinical diagnostic model to predict colonoscopy insertion time and identify difficult colonoscopy patients.

DETAILED DESCRIPTION:
The cecal intubation time (CIT) refers to the time required for the tip of the colonoscope to reach the cecum from passing through the anus. A prolonged CIT is considered a marker of difficulty in colonoscopy. A CIT greater than 10 minutes is considered a difficult colonoscopy. A longer CIT is associated with a lower adenoma detection rate, as it is an indicator of an ineffective colonoscopy, while a shorter CIT will provide the endoscopist with more time for colonoscope retrieval, increasing the likelihood of adenoma detection.

Research has identified factors that influence CIT, including age, gender, body mass index (BMI), waist circumference, bowel preparation, and prior abdominal surgery history.

Personality traits have been found to be associated with the onset of many diseases, such as hypertension and A-type personality, depression, and neurotic personality. According to the Big Five personality theory, personality can be decomposed into five dimensions: openness (O), conscientiousness (C), extraversion (E), agreeableness (A), and neuroticism (N). The Big Five personality theory is a commonly used personality typology in scientific research and has been confirmed in numerous studies. The Big Five Personality Inventory (BFI) is a tool for detecting the classification of the Big Five personality traits. The Chinese version of the Big Five Personality Inventory and norms were jointly revised by Professor Li Jian from the Department of Psychology, Beijing Normal University, and the scale norms were constructed to include people of different age groups. The scale has shown excellent reliability and validity.

The discovery of the brain-gut axis suggests that neural activity can affect the intestinal activity in various ways directly or indirectly, thereby affecting the difficulty of colonoscopy, but there is still a lack of research on the relationship between personality types and difficult colonoscopy, and the specific correlation has not been clarified. What's more important is that previous studies often used ordinary least squares regression (OLS regression) or logistic regression The purpose of this study is to investigate whether personality, BMI, age, gender, anxiety and depression index, metabolic diseases, and history of abdominal and pelvic surgery are associated with prolonged colonoscopy insertion time and difficult colonoscopy, and to construct a clinical diagnostic model by using machine learning methods to predict colonoscopy insertion time and identify difficult colonoscopy patients based on significant variables.

The basic research framework is designed as follows:

Invite patients scheduled for colonoscopy to fill out the "Personality Tendency and Colonoscopy Survey Questionnaire" before colonoscopy.

Record the completion of colonoscopy and CIT for patients during colonoscopy and record the preparation of the colon and the presence of serious organic diseases.

Collect other patient information, including age, gender, and history of major diseases.

All patients included in the study should meet the inclusion criteria and not meet the exclusion criteria.

Organize the data and divide the patients into two groups based on whether their CIT time is greater than 10 minutes.

Use t-tests and chi-square analysis to determine whether each factor is related to difficult colonoscopy, with a significance threshold of P<0.05.

Include significant variables in logistic regression for initial analysis and calculate OR.

Use LASSO regression for sparse selection and include non-zero features in the machine learning model construction.

Divide the data into training set and test set and construct random forest models, artificial neural network models, and support vector machine models, etc. Through receiver operating curve (ROC), precision, accuracy, recall rates, etc., the model's error can be evaluated, and the model's generalization ability can be compared.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy patients tested 18 to 60 years old, men and women there is no limit
* Insert the cecum complete colonoscopy examination (successfully)
* Agree and complete personality questionnaire and anxiety depression

Exclusion Criteria:

* Maternal/pregnancy/lactation
* Has a history of colorectal resection of colorectal surgery
* Have organic diseases such as severe ulcerative colitis or intestinal tumors
* Inadequate bowel preparation (bowel with feces and less than 90% visible area of mucosa)
* Confirmed with the immune system (SLE), nervous system (Alzheimer's disease), mental system (such as schizophrenia, depression), urinary system disease (CKD), and other digestive system disease
* Unable or unwilling to sign informed consent

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The study population consisted of patients who underwent colonoscopy at our hospital. They should meet the aforementioned inclusion criteria did not meet the exclusion criteria. Due to the widespread application of colonoscopy, the above patients may include patients suspected of having various organic or non-organic basic intestinal diseases, as well as health check-up patients.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of difficult colonoscopy | The evaluation of difficult colonoscopies was performed immediately after the patient completed the questionnaire at the next colonoscopy
  CIT(cecum insertion time) was applied to evaluate difficult colonoscopy, a prolonged CIT (>10min) was considered difficult colonoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Center MM, Jemal A, Smith RA, Ward E. Worldwide variations in colorectal cancer. CA Cancer J Clin. 2009 Nov-Dec;59(6):366-78. doi: 10.3322/caac.20038. PMID 19897840
- [Background] Brenner H, Chang-Claude J, Rickert A, Seiler CM, Hoffmeister M. Risk of colorectal cancer after detection and removal of adenomas at colonoscopy: population-based case-control study. J Clin Oncol. 2012 Aug 20;30(24):2969-76. doi: 10.1200/JCO.2011.41.3377. Epub 2012 Jul 23. PMID 22826281
- [Background] Jaruvongvanich V, Sempokuya T, Laoveeravat P, Ungprasert P. Risk factors associated with longer cecal intubation time: a systematic review and meta-analysis. Int J Colorectal Dis. 2018 Apr;33(4):359-365. doi: 10.1007/s00384-018-3014-x. Epub 2018 Mar 9. PMID 29520457
- [Background] Terracciano A. The Italian version of the NEO PI-R: Conceptual and empirical support for the use of targeted rotation. Pers Individ Dif. 2003;35(8):1859-1872. doi: 10.1016/S0191-8869(03)00035-7. PMID 19002272
- [Background] Zhang B, Li YM, Li J, Luo J, Ye Y, Yin L, Chen Z, Soto CJ, John OP. The Big Five Inventory-2 in China: A Comprehensive Psychometric Evaluation in Four Diverse Samples. Assessment. 2022 Sep;29(6):1262-1284. doi: 10.1177/10731911211008245. Epub 2021 Apr 22. PMID 33884926